CLINICAL TRIAL: NCT03641976
Title: A Randomized, Open-label, Multicenter Phase II Study of Bevacizumab, Infusional Fluorouracil, Leucovorin, Oxaliplatin, and Irinotecan (A-FOLFOXIRI) Compared With Bevacizumab, Infusional Fluorouracil, Leucovorin, and Irinotecan/Oxaliplatin (A-FOLFIRI/FOLFOX) as First-line Treatment for Metastatic Right-sided Colon Cancer
Brief Title: A Study of Bevacizumab, Infusional Fluorouracil, Leucovorin, Oxaliplatin, and Irinotecan (A-FOLFOXIRI) Compared With Bevacizumab, Infusional Fluorouracil, Leucovorin, and Irinotecan/Oxaliplatin (A-FOLFIRI/FOLFOX) as First-line Treatment for Metastatic Right-sided Colon Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0460
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Unresectable Metastatic Right-sided Colon Cancer Starting First-line Combination Chemotherapy; Unresectable Metastatic Right-sided Colon Cancer, Stage IV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (A-FOLFOXIRI) (Experimental): Patients receive irinotecan hydrochloride IV over 1 hour, oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and bevacizumab IV on day 1. Patients also receive fluorouracil IV continuously over 48 hours beginning on day 1.
  Interventions: Drug: A-FOLFOXIRI
- Arm II (A-FOLFOX/A-FOLFIRI) (Active Comparator): Patients receive irinotecan hydrochloride IV over 1 hour (or oxaliplatin IV over 2 hours), leucovorin calcium IV over 2 hours, fluorouracil IV bolus, and bevacizumab IV on day 1. Patients also receive fluorouracil IV continuously over 48 hours beginning on day 1.
  Interventions: Drug: Arm II (A-FOLFOX/A-FOLFIRI)

INTERVENTIONS:
Drug: A-FOLFOXIRI — Arm I (A-FOLFOXIRI)
  Biological: bevacizumab Given IV
  Drug: fluorouracil Given IV
  Drug: irinotecan hydrochloride Given IV
  Drug: leucovorin calcium Given IV
  Drug: oxaliplatin Given IV
  Arms: Arm I (A-FOLFOXIRI)
Drug: Arm II (A-FOLFOX/A-FOLFIRI) — Arm II (A-FOLFOX/A-FOLFIRI)
  Biological: bevacizumab Given IV
  Drug: fluorouracil Given IV
  Drug: irinotecan hydrochloride Given IV
  Drug: leucovorin calcium Given IV
  Arms: Arm II (A-FOLFOX/A-FOLFIRI)

SUMMARY:
RATIONALE: Recently, the importance of prognosis according to the location of the primary tumor in colorectal cancer has been raised. In the CALGB / SWOG 80405 study published in 2016, the addition of bevacizumab or cetuximab to the first line FOLFIRI / FOLFOX in KRAS (codon 12, 13) wild type metastatic colorectal cancer (mCRC) patients did not show a significant difference between overall survival (OS) and progression free survival (PFS) in both groups. Alan P. Venook et al. published a follow-up subgroup analysis on the effect of primary tumor location at 2016 ASCO. In the treatment group with cetuximab, the difference in treatment effect was significant according to the primary tumor location. The right colon cancer showed a poor prognosis for cetuximab treatment. (PFS: 7.8 vs 12.4 months, HR 1.56, p <0.0001 / OS: 16.7 vs 36.0months, HR 1.87, P <0.0001).

Therefore, the investigators propose a phase II trial for the efficacy evaluation of bevacizumab-FOLFOXIRI and bevacizumab-FOLFIRI or FOLFOX treatment in patients with poor prognosis of unresectable right-sided colorectal cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a multicenter study. Patients are stratified according to ECOG performance status (0 vs 1-2), prior adjuvant chemotherapy (yes vs no), and participating center. Patients are randomized to 1 of 2 treatment arms.

Arm I (A-FOLFOXIRI): Patients receive irinotecan hydrochloride IV over 1 hour, oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and bevacizumab IV on day 1. Patients also receive fluorouracil IV continuously over 48 hours beginning on day 1.

Arm II (A-FOLFOX/FOLFIRI): Patients receive irinotecan hydrochloride IV over 1 hour (or oxaliplatin IV over 2 hours), leucovorin calcium IV over 2 hours, fluorouracil IV bolus, and bevacizumab IV on day 1. Patients also receive fluorouracil IV continuously over 48 hours beginning on day 1.

In both arms, treatment repeats every 2 weeks for up to 12 courses. After the 12 cycle treatment finished, investigator decides whether to keep the study drug. Treatment continues in the absence of disease progression, withdrawal consent, or unacceptable toxicity. If treatment with oxaliplatin or irinotecan is difficult due to side effects, treatment with bevacizumab, fluorouracil, and leucovorin calcium continues in the absence of disease progression, withdrawal consent, or unacceptable toxicity.

Patients undergo serum extraction and blood sample collection periodically for genomic, ctDNA and translational study. Patients also undergo collection of tumoral sections from paraffin embedded primary and/or metastatic lesions periodically for immunohistochemical analyses.

After completion of study treatment, patients are followed every 6 months for survival and other treatments.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of unresectable recurrent or advanced stage IV right-sided colon cancer (The definition of the right colon cancer is confirmed by the colonoscopy result, the surgical report, or the image reading paper including CT, MRI, and PET CT. (cecum~splenic flexure))
* Not previously treated with chemotherapy for metastatic disease
* At least one measurable lesion according to RECIST criteria
* Age over 19 years old
* ECOG 0~2
* Life expectancy of at least 3 months
* Adequate major organ functions
* ANC ≥ 1.5 x 109/L
* PLT ≥ 100 x 109/L
* Hb ≥ 9.0 g/dL (can be corrected by blood transfusion)
* Total bilirubin ≤ upper normal limit(UNL) * 1.5
* ALT , AST ≤ UNL * 3 (in case of liver metastasis, ALT , AST ≤ UNL * 5), alkaline phosphatase ≤ UNL *3 (in case of liver metastasis, ALP ≤ UNL * 5
* adequate renal function : corrected creatinine clearance by Cockcroft and Gault formula ≥ 30mL/min
* Urine dipstick of proteinuria <2+. Patients discovered to have 2+ proteinuria on dipstick urinalysis at baseline, should undergo a 24-hour urine collection and must demonstrate 1 g of protein/24 hr.
* Written informed consent.

Exclusion Criteria:

* Previously treated with chemotherapy for metastatic disease
* Within 6 months after adjuvant chemotherapy
* Major surgical procedure within 28 days prior to study treatment start, or patients who have not fully recovered from major surgery
* Radiotherapy to target lesion within 4 weeks before the study (A 2-week washout is permitted for palliative radiation.)
* Has known uncontrolled active CNS metastases and/or carcinomatous meningitis
* Peripheral neuropathy CTCAE v4.03 ≥ grade 2
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

Note: Participants with basal cell carcinoma of skin, squamous cell carcinoma of the skin, low grade thyroid cancer or carcinoma in situ (eg, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.

* Has an active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy, such as thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, is not considered a form of systemic systemic treatment and is allowed.
* Uncontrolled hypertension or clinically active cardiovascular disease: for example, cerebrovascular accident or transient ischemic attack, unstable angina, myocardial infarction within 24 weeks prior to randomization. Have symptomatic congestive heart failure (CHF; New York Heart Association II-IV) or symptomatic or poorly controlled cardiac arrhythmia.
* Have significant bleeding disorders, or evidence of bleeding diathesis or coagulopathy
* Have had a significant bleeding episode from the gastrointestinal (GI) tract or lung
* Have a history of GI perforation and/or fistula, or intra-abdominal abscess within 24 weeks prior to randomization.
* Have a history of HNPCC syndrome or polyposis
* Have experienced any arterial thromboembolic event or ongoing treatment with anticoagulants for therapeutic purpose within 24 weeks prior to randomization.
* Has a known history of human immunodeficiency virus (HIV) infection
* Are pregnant or breast feeding. Females of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to first dose of study treatment. For women of childbearing potential and men, agreement to remain abstinent or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 30 days after the last dose of study drugs. Postmenopausal women is defined that : 1) must have been amenorrheic for at least 12 months, > 50 years old or 2) Age ≤ 50 years old and amenorrheic for 12 or more months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression and follicle-stimulating hormone (FSH) and estradiol in the postmenopausal range (>40 mIU/mL), 3) prior bilateral oophorectomy
* Patients who are hypersensitive reaction to experimental drugs
* Patients who are hypersensitive to CHO cell products or other recombinant or humanized antibodies
* In case of contraindication of experimental drugs
* Have any condition (eg, psychological, geographical, or medical) that does not permit compliance with the study and follow-up procedures or suggest that the patient is, in the investigator's opinion, not an appropriate candidate for the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
6-month PFS rate (%) | 6 months
  To compare the 6-month progression free survival (PFS) rate (%) of bevacizumab in combination with oxaliplatin, irinotecan and infusional 5FU/LV (A-FOLFOXIRI regimen) to bevacizumab in combination with oxaliplatin or irinotecan and infusional 5FU/LV (A-FOLFOX/A-FOLFIRI regimen) in not previously treated, unresectable stage IV right-sided colon cancer

SECONDARY OUTCOMES:
overall survival(OS) | 4 years
  To compare the overall survival (OS) between treatment arms
progression free survival(PFS) | 4 years
  To compare the progression free survival (PFS) between treatment arms
adverse events | 4 years
  To evaluate the safety profile including long-term adverse events between treatment arms
surrogate markers predictive of survival: ctDNA | 4 years
  To evaluate the correlation between 6-month PFS rate(%) and change in ctDNA

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Cancer Center, Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided